CLINICAL TRIAL: NCT05829356
Title: A Phase I, Parallel, Randomized, Active-controlled, Multi-center, Dose-escalation Study With Early Safety Data Reviews to Assess Safety and Immunogenicity of One Monovalent Modified Influenza mRNA Vaccine Encapsulated in LNP, in Adults Aged 18 to 49 Years and 60 Years and Above.
Brief Title: Substudy 01 - Safety and Immunogenicity of One Monovalent Modified mRNA Vaccine Encoding Influenza Hemagglutinin With LNP, in Adult Participants Aged 18 to 49 Years and 60 Years and Above
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VAV00019; U1111-1278-3835 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-04-06; First posted 2023-04-25 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Influenza Immunization
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This study will be blinded to participants and sites (except for those preparing/administering study interventions. The sponsor will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1: H3 mRNA /LNP dose 1 (Experimental): Participants will receive one intramuscular (IM) dose of H3 mRNA/LNP at Day 01
  Interventions: Biological: H3 mRNA / LNP Vaccine
- Group 2: H3 mRNA /LNP dose 2 (Experimental): Participants will receive one IM dose of H3 mRNA/LNP at Day 01
  Interventions: Biological: H3 mRNA / LNP Vaccine
- Group 3: H3 mRNA /LNP dose 3 (Experimental): Participants will receive one IM dose of H3 mRNA/LNP at Day 01
  Interventions: Biological: H3 mRNA / LNP Vaccine
- Group 4: H3 mRNA /LNP dose 4 (Experimental): Participants will receive one IM dose of H3 mRNA/LNP at Day 01
  Interventions: Biological: H3 mRNA / LNP Vaccine
- Group 5: H3 mRNA /LNP dose 5 (Experimental): Participants will receive one IM dose of H3 mRNA/LNP at Day 01
  Interventions: Biological: H3 mRNA / LNP Vaccine
- Group 6 (Control Group): RIV4 dose (Active Comparator): Participants will receive one IM dose of RIV4 at Day 01
  Interventions: Biological: Quadrivalent recombinant influenza Vaccine (RIV4)

INTERVENTIONS:
Biological: H3 mRNA / LNP Vaccine — Pharmaceutical Form: Suspension for injection
  Route of Administration: Intra-Muscular
  Arms: Group 1: H3 mRNA /LNP dose 1; Group 2: H3 mRNA /LNP dose 2; Group 3: H3 mRNA /LNP dose 3; Group 4: H3 mRNA /LNP dose 4; Group 5: H3 mRNA /LNP dose 5
Biological: Quadrivalent recombinant influenza Vaccine (RIV4) — Pharmaceutical Form: Solution for injection in a pre-filled syringe
  Route of Administration: Intra-Muscular
  Other Names: Flublok Quadravalent®
  Arms: Group 6 (Control Group): RIV4 dose

SUMMARY:
This is a Phase 1, parallel, randomized, active-controlled, multi-center, dose-esclation study with a Master Protocol design which will include several substudies that are developed to evaluate the safety and immunogenicity of different dose levels of modified messenger ribonucleic acid (mRNA) vaccines encoding full length hemagglutinin (HA) sequence of influenza virus encapsulated in lipid nanoparticles (LNPs) (hereafter referred to as HA mRNA vaccines) compared to control(s). The HA mRNA vaccine candidates and control(s) are presented in the substudy protocols.

The aim is to generate clinical data across different substudies to provide learnings regarding the mRNA technology to support optimization of the mRNA platform including mRNA and LNP design and to support the decision of LNP and dose selection for future projects using mRNA technology.

The purpose of this Substudy 01 is to evaluate the safety and immunogenicity of a single IM injection of up to 5 dose levels of a monovalent modified mRNA encoding the full-length HA sequence of A/Tasmania/503/2020 (H3N2) influenza virus encapsulated in LNP (hereafter referred to as H3 mRNA /LNP) administered as a single intramuscular (IM) injection in adults 18 to 49 years of age and 60 years of age and above, compared to the following active control: a quadrivalent recombinant influenza vaccine (RIV4).

DETAILED DESCRIPTION:
The study duration per participant will be approximately 6 months with 1 injection of one of the different HA mRNA vaccines or control for each substudy and a dose-escalation with sequential enrollment (sentinel cohort followed by main cohort).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above on the day of inclusion

  *Aged 18 years to 49 years or 60 years and above on the day of inclusion (substudy 01)
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

  * Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be postmenopausal for at least 1 year, or surgically sterile.

OR

• Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to study intervention administration until at least 12 weeks after study intervention administration.

* A female participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) at the screening visit.
* Inclusion Criteria to be Checked at Visit 1 (Day 1)

Participants are eligible for the study only if all of the following criteria are met:

A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

• Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be postmenopausal for at least 1 year, or surgically sterile.

OR

• Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to study intervention administration until at least 12 weeks after study intervention administration.

A female participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) within 8 hours before the first dose of study intervention.

Exclusion Criteria:

* Previous vaccination against influenza in the previous 6 months with an investigational or marketed vaccine
* Any screening laboratory parameter with laboratory abnormalities that are greater than Grade 1 or deemed clinically significant in the opinion of the Investigator

  * OR, any screening Liver Function Test (ALT, AST, Bilirubin) > 1.2x Upper Limit of Normal or any other screening laboratory parameter outside of the range of normal limits for age and gender
* Positive test for human immunodeficiency virus (HIV) antigen and/or antibodies (Abs), hepatitis B (HB) virus surface antigen (HBsAg), hepatitis B core antibodies (HBcAb), or hepatitis C virus antibodies (HCV Abs)
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the study intervention components (eg, polyethylene glycol [PEG], polysorbate); history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances; any allergic reaction (eg, anaphylaxis) after administration of mRNA COVID-19 vaccine
* Previous history of myocarditis, pericarditis, and/or myopericarditis
* Screening electrocardiogram (ECG) or troponin value that is consistent with probable or possible myocarditis, pericarditis, and/or myopericarditis or screening ECG that demonstrates clinically relevant abnormalities that may affect participant safety or study results
* Self-reported thrombocytopenia, contraindicating intramuscular vaccination based on Investigator's judgment
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination based on Investigator's judgment
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with study conduct or completion
* Alcohol, prescription drug, or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion
* Receipt of any vaccine in the 4 weeks preceding study enrollment or planned receipt of any vaccine in the 4 weeks following study intervention administration
* Receipt of any mRNA vaccine/product in the 2 months preceding study enrollment or planned receipt of any mRNA vaccine/product within the 2 months following study intervention administration
* Receipt of immune globulins, blood or blood-derived products in the past 3 months -Participation at the time of study enrollment (or in the 4 weeks preceding study enrollment or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure
* Previous vaccination against influenza in the previous 6 months with an investigational or marketed vaccine
* Exclusion criteria to be checked at Visit 1 Day 1:

  * Moderate or severe acute illness/infection (according to Investigator's judgment) or febrile illness (temperature ≥ 38.0°C [100.4°F]) on the day of vaccination. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with immediate adverse events (AEs) | Within 30 minutes after vaccination
  Unsolicited systemic AEs that occur within 30 minutes after vaccination
Number of participants with solicited injection site or systemic reaction | Within 7 days from vaccination
  Number of participants reporting Adverse reactions pre-listed in the protocol and case report form (CRF)
  * Injection site reactions: pain, redness, swelling
  * Systemic reactions: fever, headache, malaise, myalgia, arthralgia, chills
Number of participants with unsolicited adverse events | Up to 28 days after injection
  Unsolicited (spontaneously reported) adverse events not fulfilling criteria for solicited reactions
Presence of out-of-range biological test results | At Day 3, Day 9 or Day 29
  Number of participants with biological safety assessment values out of normal range (as per the laboratory performing the test)
Presence of serious adverse events (SAEs) | Throughout Study (up to approximately Month 6)
  Number of participants experiencing SAEs
Presence of adverse events of special interest (AESIs) | Throughout Study (up to approximately Month 6)
  Number of participants experiencing AESIs
Hemagglutination inhibition (HAI) antibody (Ab) response to homologous strain | Day 29
  Antibody are expressed as geometric mean titers (GMTs) at baseline and post-baseline
HAI titers at D01 | Day 1
  Antibody titers are expressed as GMTs at baseline and post-baseline
HAI titers at D29 | Day 29
  Antibody titers are expressed as GMTs at baseline and post-baseline
Individual HAI Ab titer ratio | Day 1 through Day 29
  Individual HAI Ab titer ratio will be calculated as: D29/D01
Number of Participants with Vaccine Response or Seroconversion | Day 1 through Day 29
  Seroconversion (HAI Ab titer < 10 [1/dil] at D01 and post-injection titer ≥ 40 [1/dil] at D29, or titer ≥ 10 [1/dil] at D01 and a ≥ 4-fold increase in titer [1/dil] at D29)
2-fold and 4-fold rise in HAI titers from D01 to D29 | Day 1 to Day 29
  Expressed as percentage post-baseline
Percentage of participants with detectable antibody HAI titers greater than or equal to (≥) 40 [1/dil] | Day 29
Geometric Mean Titers (GMTs) of neutralizing antibody (nAb) titers at Day 1 | Day 1
  Nab titers at Day 1
Geometric Mean Titers (GMTs) of neutralizing antibody (nAb) titers at Day 29 | Day 29
  Nab titers at Day 29
Individual nab titer ratio | Day 1 through Day 29
  Individual nab titer ratio will be calculated as: D29/D01
2-fold and 4-fold increase in neutralizing Ab titers from D01 to D29 | Day 1 to Day 29
  Expressed as percentage post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (8):
- Australia (4):
  - Investigational Site Number : 0360004, Herston, Queensland
  - Investigational Site Number : 0360001, Morayfield, Queensland
  - Investigational Site Number : 0360002, Camberwell, Victoria
  - Investigational Site Number : 0360003, Adelaide
- United Kingdom (4):
  - Investigational Site Number : 8260002, Leicester, Leicestershire
  - Investigational Site Number : 8260001, London, London, City of
  - Investigational Site Number : 8260004, London, London, City of
  - Investigational Site Number : 8260003, Sheffield, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VAV00019 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25377&tenant=MT_SNY_9011